CLINICAL TRIAL: NCT05406596
Title: LiquID Guide Catheter Extension Safety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seigla Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200-0004
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- LiquID GCE Use (Experimental)
  Interventions: Device: LiquID GCE Use

INTERVENTIONS:
Device: LiquID GCE Use — Use of the LiquID GCE to aid in percutaneous coronary intervention (PCI)

SUMMARY:
Single arm, open label, historically controlled, multicenter study evaluating the primary safety and performance of the LiquID Guide Catheter Extension

DETAILED DESCRIPTION:
The study will consist of evaluating the safety and performance of the LiquID Guide Catheter Extension (GCE) compared to historical data. The safety measures will consist of procedural Major Adverse Cardiac Events (MACE) while performance measures will include Device Oriented Clinical Outcomes.

ELIGIBILITY:
Inclusion Criteria - participants must be:

1. scheduled for non-emergent, percutaneous coronary procedure in which the use of a guide catheter extension is anticipated
2. able to provide informed consent to participate in the study

Exclusion Criteria - participants must not have:

1. evidence of ongoing ST-elevation myocardial infarction (STEMI) or STEMI treatment for late presentation STEMI with index admission (stabilized acute coronary syndrome allowed)
2. left ventricular ejection fraction <20%
3. required intervention in a saphenous vein graft
4. an intolerance or known allergy to medications/contrast expected to be used during the procedure or during hospital stay
5. had a cardiac intervention within two weeks of the procedure
6. renal insufficiency (serum creatinine of > 2.3 mg/dl)
7. active gastrointestinal bleeding
8. an active infection or fever (>37.8º C) that may be due to infection
9. significant anemia (hemoglobin < 8.0 mg / dl)
10. severe uncontrolled systemic hypertension (systolic press. > 240 mm Hg within the past month)
11. a severe electrolyte imbalance
12. congestive heart failure (NYHA Class IV)
13. presented with an acute coronary syndrome where serum troponin concentrations have not been demonstrated to be declining prior to the scheduled procedure (within the past two weeks)
14. uncontrolled diabetes (> 2 serum glucose concentrations of > 350 mg/dl within the past 7 days)
15. participation in an investigational protocol
16. unwillingness or inability to comply with any protocol requirements
17. angina, or ischemia caused by occluded artery
18. other clinical conditions, that in the opinion of the investigator significantly compromise the ability to perform a safe and/or effective procedure

Vulnerable Population Exclusion - participants must not be:

1. under 18 years old
2. pregnant or nursing
3. immuno-compromised
4. over 89 years old
5. incapacitated, mentally compromised or otherwise incapable of understanding and/or providing informed consent (including emergency situations)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Henriksen, BSc, MB ChB, PhD, FRCP, Principal Investigator — Royal Edinburgh
Locations (8):
- Ziekenhuis Oost-Limburg, Genk, Belgium
- Ireland (3):
  - Mater Private, Cork
  - Mater Private, Dublin
  - Galway University Hospital, Galway
- United Kingdom (4):
  - University Hospitals Bristol, Bristol
  - Royal Edinburgh, Edinburgh
  - Golden Jubilee, Glasgow
  - St. George's Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LiquID GCE Use
Started | 86
Completed | 86
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who were successfully screened
Arm/Group | LiquID GCE Use
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 36
  Belgium | 19
  Ireland | 31
Diabetes [Count of Participants; unit: Participants] | 20
Hypertension [Count of Participants; unit: Participants] | 57
Hypercholesterolemia [Count of Participants; unit: Participants] | 68
Medication Allergy [Count of Participants; unit: Participants] | 13
Infectious Disease (HIV, TB, etc.) [Count of Participants; unit: Participants] | 2
History of CABG [Count of Participants; unit: Participants] | 11
History of PCI [Count of Participants; unit: Participants] | 41
History of Angiography (no PCI) [Count of Participants; unit: Participants] | 46
History of Peripheral PTA [Count of Participants; unit: Participants] | 4
History of Cerebrovascular PTA [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With In-hospital Major Adverse Cardiac Events (MACE)
Description: * Device-caused events including:
    * Target vessel dissection
    * Longitudinal stent deformation
    * Proximal collar stent stripping
  * Cardiac death
  * Stroke
  * Peri-procedural myocardial infarction (MI) based on participant symptoms, ECG changes and/or SCAI definition (if cardiac enzymes are available)
Time Frame: 48 hours or discharge (whichever comes first)
Population: All participants were analyzed for any adverse events that may have occurred.
Measure: Count of Participants; unit: Participants
Arm/Group | LiquID GCE Use
Number analyzed (Participants) | 86
Participants | 2

2. Secondary Outcome: The Number of Participants With Device Oriented Clinical Outcome
Description: Successful deployment and retrieval of the LiquID device without any device deficiencies or where use of the LiquID device directly leads to a MACE, target vessel dissection, longitudinal stent deformation or proximal collar stent stripping.
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | LiquID GCE Use
Number analyzed (Participants) | 86
Participants | 79

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | LiquID GCE Use
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 4/86
Other Adverse Events (participants affected / at risk) | 15/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LiquID GCE Use (N=86)
Dissection (Vascular disorders) | 1 (1)
Dissection/MI (Vascular disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Palpitations, dizziness (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LiquID GCE Use (N=86)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Arm Wound (Injury, poisoning and procedural complications) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3)
Chest Pain (Injury, poisoning and procedural complications) | 1 (1)
Chest Pain (General disorders) | 3 (3)
Left Foot Swelling (Vascular disorders) | 1 (1)
Transient Ischemic Attack (Cardiac disorders) | 1 (1)
Orthostatic hypotension (Blood and lymphatic system disorders) | 1 (1)
Left Arm Cramping (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT05406596/Prot_SAP_000.pdf